CLINICAL TRIAL: NCT01845766
Title: Effects of Early Exercise Rehabilitation on Long-term Functional Recovery in Patients With Severe Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4-2012-0710
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Severe Sepsis or Septic Shock
Keywords: sepsis, septic shock, rehabilitation, exercise
MeSH Terms: conditions — Sepsis; Shock, Septic; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rehabilitation arm (Experimental): daily standardized exercise rehabilitation during the admission period, and daily standardized self exercise after discharge
  Interventions: Other: exercise rehabilitation
- control arm (No Intervention)

INTERVENTIONS:
Other: exercise rehabilitation
  Arms: rehabilitation arm

SUMMARY:
We hypothesized that early exercise rehabilitation for patients with severe sepsis or septic shock would decrease their functional disability and cognitive impairment. We plan to enroll patients with severe sepsis and septic shock who admitted an urban teaching hospital in Seoul, South Korea via ER. We will randomize those subjects into the intervention group which will take a standardized rehabilitation with routine clinical care for sepsis and the control group which will take routine clinical care for sepsis. And, we plan to assess their functional activity using ADL, IADL and SF-36, and cognitive function using MMSE at the time of enrollment, 28 days, and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥20;
2. confirmed or suspected infection;
3. two or more among 1)-4) 1) body temperature >38˚C or <36˚C 2) heart rate >90/min 3) respiratory rate >20/min or PaCO2<32 mmHg 4) WBC >12000/mm3, <4000/mm3, or band forms >10%;
4. within 48 hours after arriving ER

Exclusion Criteria:

1. severe functional disability before admission;
2. central nervous system infection;
3. contraindication for exercise rehabilitation according to the investigators' decision;
4. severe medical illness or mental problem or laboratory abnormality which can confound the results;
5. pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Severe functional disability | 6 months after enrollment
  We will assess the functional activity with 0-11 score of 6 ADL(walking, dressing, bathing, eating, getting into and out of bed, toileting) and 5 IADL(preparing a hot meal, shopping for groceries, making telephone calls, taking medicines, managing money). If the patient has a score 4 or more, the patient will be considered to have a severe functional disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, Seoul, South Korea